CLINICAL TRIAL: NCT03291444
Title: A Clinical Study of Chimeric Antigen Receptor T Cells Combined With Eps8 Peptide Specific Dendritic Cell for Patients With Relapsed/Refractory Leukemia and Myelodysplastic Syndromes
Brief Title: CAR-T Cells Combined With Peptide Specific Dendritic Cell in Relapsed/Refractory Leukemia/MDS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: Shenzhen Geno-Immune Medical Institute (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-XYNK-001
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Leukemia, Acute Lymphocytic (ALL); Leukemia, Acute Myelogenous (AML); Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAR-T cells combined with peptide specific dendritic cell (Experimental): CAR-T cells combined with Eps8 peptide specific dendritic cell,or CAR-T cells combined with WT1 peptide specific dendritic cell
  Interventions: Biological: Chimeric antigen receptor T cells; Biological: peptide specific dendritic cell
- Chimeric antigen receptor T cells (Active Comparator): After pretreatment, chimeric antigen receptor T cells will be transfused.
  Interventions: Biological: Chimeric antigen receptor T cells

INTERVENTIONS:
Biological: Chimeric antigen receptor T cells — After pretreatment, chimeric antigen receptor T cells will be transfused.
  Other Names: CAR-T
Biological: peptide specific dendritic cell — After transfusion of chimeric antigen receptor T cells, Eps8 or WT1 peptide specific dendritic cell were intradermal injected.
  Other Names: WT1 peptide specific dendritic cell; Eps8 peptide specific dendritic cell
  Arms: CAR-T cells combined with peptide specific dendritic cell

SUMMARY:
The main purpose of this study is to verify the safety and potential effectiveness of CART cells combined with peptide specific dendritic cell in relapsed/refractory leukemia.

DETAILED DESCRIPTION:
A prospective study to evaluate the safety and efficacy of Chimeric antigen receptor T cells combined with Eps8 or WT1（Wilms tumor 1） peptide specific dendritic cell for patients with relapsed/refractory leukemia. There are options for CAR-targets: CD19, CD20, CD22 and CD10 for acute lymphoblastic leukemia; CD33, CD38 CD56, CD117, CD123, CD34 and Muc1 for acute myeloid leukemia and Myelodysplastic Syndrome. Progression free survival, overall Survival, overall response rate, and duration of response were monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor type: Acute Myeloid Leukemia (AML) and Acute Lymphoblastic Leukemia (ALL) according to the WHO criteria (at least 20% blasts in the marrow). All FAB subtypes except M3. Patients with Myelodysplastic Syndrome, category of Refractory Anemia with Excess Blasts (RAEB): RAEB I (WHO: medullary blast count ≤ 10% and a peripheral blast count ≤ 5%) and RAEB II (WHO: medullary blast count > 10% and/or > 5% peripheral blasts) can be included in the study in absence of other non-experimental treatment modalities.
2. Positive antigen for any of CD19, CD20, CD22, CD10, CD33, CD38, CD56, CD117, CD123, CD34, or Muc1.Simultaneously ,high expression of EPS8 or WT1 in acute leukemia.
3. Relapsed/Refractory leukemia patients：

   * Did not achieve complete remission after 2 times of standard plan chemotherapy.
   * Relapsed after first induction chemotherapy.
   * Did not response to chemotherapy before HSCT or relapsed after HSCT.
   * Cannot receive allo-HSCT or refuse to receive allo-HSCT.
   * Relapsed after CAR-T cell infusion.
4. Age greater than 18 year and less than 80 years.
5. Objectively assessable parameters of life expectancy: more than 3 months.
6. Performance status: WHO PS grade 0-1 (ECOG performance status 0 or 1).
7. Meet the following criteria for apheresis：WBC >= 3,000/L, Hb >= 8.0 g/dL, platelet count >= 80,000/mm3, <= 600,000/mm3.
8. Pulmonary function: Peripheral blood oxygen saturation greater than 90%; Cardiac function: Left ventricular ejection fraction >60%.
9. Prior and concomitant associated diseases allowed with the exception of underlying autoimmune disease and positive serology for HIV/HBV/HCV.
10. No concomitant use of immunosuppressive drugs.
11. Adequate renal and liver function, i.e. creatinin, bilirubin, and aminotransferase =< 1.2 times the upper limit of normal.
12. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
13. Women of child-bearing potential should use adequate contraception prior to study entry and for the duration of study participation.
14. Written informed consent obtained.

Exclusion Criteria:

1. Patients with severe complications: cardiovascular disorders, respiratory disorders, renal dysfunction, immunodeficiency, hematological disorders, autoimmune diseases, sever allergy and severe infectious disease.
2. Patients who should receive systemic administration of steroid or immunosuppressive agents.
3. Presence of active brain metastases.
4. Pregnant, lactating, or possibly pregnant women, or willing to be pregnant.
5. Severe psychiatric disorder.
6. Active multiple cancers.
7. Patients have received other genetic therapy products.
8. Transfection efficiency was less than 30%.
9. Inappropriate for study entry judged by an attending physician.
10. patients who have sensitivity to drugs that provide local anesthesia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events, according to NCI CTCAE Version 4.0 | up to 12 months
  Incidence and severity of cytokine release syndrome(CRS): The systemic inflammatory response in patients with significantly increased IL-6 and other cytokines during the observation period is defined as CRS, which is divided into 1-5 grades, 1-2 Grade is mild, grade 3-5 is severe

SECONDARY OUTCOMES:
Progression free survival time | 2 years
  Time from random to the first occurrence of disease progression.
Overall survival time | 2 years
  Time from randomization to death due to any cause
Overall response rate | 2 years
  The proportion of the total number of patients with complete remission and partial remission (CR+PR) after treatment in the total number of evaluable cases
Duration of response | 2 years
  During the observation period, the time between complete remission of bone marrow (the ratio of bone marrow blast cells is less than 5%) to the recurrence of bone marrow (the ratio of bone marrow blast cells is greater than 5%) is the continuous remission time.

CONTACTS AND LOCATIONS:
Overall Officials: Yuhua Li, M.D, Ph.D, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tu S, Zhou L, Huang R, Zhou X, Yang J, He Y, Hu Y, Zhang H, Xie X, Li Y. Dendritic cell vaccines extend CAR T-cell persistence and improve the efficacy of CD19 CAR T-cell therapy in refractory or relapsed adult B-ALL patients. Am J Hematol. 2024 Jul;99(7):1437-1440. doi: 10.1002/ajh.27349. Epub 2024 May 7. No abstract available. PMID 38712616